CLINICAL TRIAL: NCT06002763
Title: Evaluation of Patient-Reported Outcomes Measurement Information System (PROMIS)-29 v2.1 for Postpartum Women
Status: Recruiting | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 23-03
Record Dates: First submitted 2023-08-16; First posted 2023-08-21 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Well-Being, Psychological
Keywords: cesarean delivery; vaginal delivery; postpartum recovery
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Vaginal delivery: Patients who have vaginal deliveries with neuraxial labour analgesia.
  Interventions: Other: PROMIS-29 v2.1 (Patient-Reported Outcomes Measurement Information System); Other: WHOQoLBREF (World Health Organization Quality of Life Brief Version); Other: EQ-5D-3L1 (not an acronym)
- Cesarean delivery: Patients who have a scheduled cesarean delivery with neuraxial anesthesia.
  Interventions: Other: PROMIS-29 v2.1 (Patient-Reported Outcomes Measurement Information System); Other: WHOQoLBREF (World Health Organization Quality of Life Brief Version); Other: EQ-5D-3L1 (not an acronym)

INTERVENTIONS:
Other: PROMIS-29 v2.1 (Patient-Reported Outcomes Measurement Information System) — PROMIS-29 is a survey designed to screen for pain, impairments in mood, physical function, and activities of daily living.
  Other Names: Patient-Reported Outcomes Measurement Information System
Other: WHOQoLBREF (World Health Organization Quality of Life Brief Version) — The WHOQOL-BREF is a 26-item version of the 100-item WHOQOL-100 quality of life measure that addresses four quality of life domains: physical health, psychological health, social relationships and environment.
  Other Names: World Health Organization Quality of Life Brief Version
Other: EQ-5D-3L1 (not an acronym) — The EQ-5D-3L1 is a generic measure of health status consisting of two parts. The first part assesses health in five dimensions: MOBILITY, SELFCARE, USUAL ACTIVITIES, PAIN / DISCOMFORT, ANXIETY/DEPRESSION. The second part of the questionnaire consists of a VAS on which the patient rates their perceived health from 0 (the worst imaginable health) to 100 (the best imaginable health).
  Other Names: Global state of health numerical rating score 1-100

SUMMARY:
There is no widely used, statistically validated assessment for physical and mental health for the short- to medium-term in a postpartum population. PROMIS-29 has been validated for the assessment of these factors in a generic population, but has not been specifically evaluated for use with postpartum women.

This study is a longitudinal, single center observational cohort study designed to evaluate the reliability of the Patient-Reported Outcomes Measurement Information System (PROMIS)-29 v2.1 survey in a postpartum population. PROMIS-29 is a survey designed to screen for pain, impairments in mood, physical function, and activities of daily living. While this survey has shown utility in other populations, it has yet to be assessed in an obstetric population. The investigators plan to recruit patients who are recently postpartum from vaginal or cesarean delivery to complete virtual surveys at defined time points (0, 2, 6, and 12 weeks after delivery). The investigators will subject survey data to statistical measures of validity and reliability comparing with contemporaneously collected surveys of established metrics for quality of life (WHOQoLBREF) and general (global) state of health (numerical rating score 1-100).

The hypothesis is that the PROMIS-29 v2.1 questionnaire is a statistically valid and reliable means of assessing physical and mental health in a postpartum population.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* singleton births
* 37 or more weeks gestational age
* multiparous or nulliparous patients
* spontaneous vaginal delivery or scheduled cesarean delivery with labor analgesia or neuraxial anesthesia
* give informed written consent

Exclusion Criteria:

* refusal to take part
* are unable to give or have withdrawn consent
* patients unable to communicate fluently in English
* patients who are less than 18 years old
* patients who had fetal demise or severely morbid fetal conditions such as intubation, cooling, expected surgical correction of congenital anomaly during hospitalization (although NICU admissions will be included)
* patients who were admitted in ICU
* patients who had failed neuraxial analgesia such as replaced epidurals or failed spinal requiring conversion to general anesthesia
* patients who had general anesthesia for cesarean delivery as defined by "GETA", including sedatives and deep sedation if not intubated
* patients who had intrapartum cesarean or had assisted/operative (i.e. vacuum, forceps) vaginal delivery.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who deliver vaginally or by scheduled cesarean section at Mount Sinai Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
PROMIS-29 v2.1 (Patient-Reported Outcomes Measurement Information System) survey score | 24 hours
  The PROMIS survey score at 24 hours postpartum
WHOQoLBREF (World Health Organization Quality of Life Brief Version) survey score | 24 hours
  The WHOQoLBREF survey score at 24 hours postpartum
EQ-5D-3L1 (not an acronym) survey score | 24 hours
  The EQ-5D-3L1 survey score at 24 hours postpartum
PROMIS-29 v2.1 (Patient-Reported Outcomes Measurement Information System) survey score | 2 weeks
  The PROMIS survey score at 2 weeks postpartum
WHOQoLBREF (World Health Organization Quality of Life Brief Version) survey score | 2 weeks
  The WHOQoLBREF survey score at 2 weeks postpartum
EQ-5D-3L1 (not an acronym) survey score | 2 weeks
  The EQ-5D-3L1 survey score at 2 weeks postpartum
PROMIS-29 v2.1 (Patient-Reported Outcomes Measurement Information System) survey score | 6 weeks
  The PROMIS survey scores at 6 weeks postpartum
WHOQoLBREF (World Health Organization Quality of Life Brief Version) survey score | 6 weeks
  The WHOQoLBREF survey score at 6 weeks postpartum
EQ-5D-3L1 (not an acronym) survey score | 6 weeks
  The EQ-5D-3L1 survey score at 6 weeks postpartum
PROMIS-29 v2.1 (Patient-Reported Outcomes Measurement Information System) survey score | 12 weeks
  The PROMIS survey score at 12 weeks postpartum
WHOQoLBREF (World Health Organization Quality of Life Brief Version) survey score | 12 weeks
  The WHOQoLBREF survey score at 12 weeks postpartum
EQ-5D-3L1 (not an acronym) survey score | 12 weeks
  The EQ-5D-3L1 survey score at 12 weeks postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Ronald George, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No